CLINICAL TRIAL: NCT04350177
Title: A Phase I, Randomized Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Determine the Safety, Tolerability and Pharmacokinetics (PK) of IkT-148009 in Older Adult and Elderly Healthy Volunteers With Extension Into Parkinson's Patients
Brief Title: A Study to Assess Single and Multiple Doses of IkT-148009 in Healthy Elderly Participants and Parkinson's Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ABLi Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: IkT-148009-101
Record Dates: First submitted 2019-12-26; First posted 2020-04-16 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2023-02

CONDITIONS: Healthy Elderly; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Sentinel dosing will be employed for each cohort in Part A, with one subject randomized to receive IkT-148009 and the other placebo on the first day. These two subjects in each cohort will be monitored for 48 hours after dosing before deciding to dose the remainder of the cohort. As such, the other six subjects in the first cohort will be dosed approximately 48 hours later. Each cohort will be monitored for at least 48 hours before deciding whether to sentinel pair in the next (higher dose) cohort, and each cohort will be dosed at approximately monthly intervals in order to allow adequate time for collection and review of safety and PK data. In Part B, 8 patients will be 3:1 randomized to placebo and dosed once per day for 7 days. In Part C, 8 patients will be 3:1 randomized to placebo and dosed once per day for 7 dayts.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (SAD) (Active Comparator): In Part A, cohorts will consist of eight (8) subjects; six (6) of whom will receive treatment with IkT-148009 and two (2) with matching placebo.
  Interventions: Drug: IkT-148009; Drug: Placebo
- Multiple Ascending Dose (MAD) (Active Comparator): In Part B, cohorts will consist of eight (8) subjects; six (6) of whom will receive treatment with IkT-148009 and two (2) with matching placebo.
  Interventions: Drug: IkT-148009; Drug: Placebo
- Multiple Ascending Dose (MAD) Parkinson's patients (Active Comparator): In Part C, cohorts will consist of eight (8) patients; six (6) of whom will receive treatment with IkT-148009 and two (2) with matching placebo.
  Interventions: Drug: IkT-148009; Drug: Placebo

INTERVENTIONS:
Drug: IkT-148009 — Oral administration gelatin capsule
Drug: Placebo — Oral administration gelatin capsule

SUMMARY:
This study investigates the safety and tolerability of drug IkT-148009 in healthy elderly volunteers (55 to 70 years old). This first-in-human study is designed in 3 parts. In Part A, healthy participants will take a single, oral dose of IkT-148009 or placebo. Part A participants will be at the study site for approximately 4 days. In Part B, healthy participants will take an oral dose of IkT-148009 once a day for 7 days. Part B participants will be at the study site for approximately 12 days. In Part C, Parkinson's patients will take an oral dose of IkT-148009 once a day for 7 days. Part C participants will be at the study site for approximately 12 days.

DETAILED DESCRIPTION:
This is a randomized, Phase 1 study in older adult or elderly healthy volunteer subjects with subsequent extension into Parkinson patients to identify the safety, tolerability, maximum tolerated dose (MTD) and the pharmacokinetic (PK) profile of IkT-148009 capsules given as single or multiple doses.

In Part A (SAD) cohorts will consist of eight (8) subjects, six (6) of whom will receive treatment with IkT-148009 and two (2) with matching placebo. Sentinel dosing will be employed on the first day of each cohort, with one subject randomized to receive IkT-148009 and the other placebo. These two subjects in each cohort will be monitored for 48 hours after dosing before deciding to dose the remainder of the cohort. The other six subjects in the first cohort will be dosed approximately 48 hours later. Each cohort will be monitored for at least 48 hours before deciding whether to administer drug to the sentinel pair for the next cohort. Each cohort will be dosed at approximately weekly intervals to allow adequate time for collection and review of safety and PK data.

A Safety Review Committee (SRC) will evaluate all available safety, tolerability, and PK data for each cohort. Escalation to a next dose will be undertaken only after these data have been reviewed by the SRC and agreement reached that it is safe to increase the dose. The SRC will not receive any unblinded PK data unless they agree to unblind a subject and/or cohort based on the completed safety review.

In Part B (MAD) cohorts will consist of eight (8) subjects, six (6) of whom will receive treatment with IkT-148009 and two (2) with matching placebo daily for up to seven consecutive days. Subjects in each cohort will be observed for 48 hours after their last dose before deciding to initiate the next (higher dose) cohort. Each cohort will be dosed at approximately weekly intervals in order to allow adequate time for collection and review of safety and PK data. At the discretion of the SRC, MAD cohorts may be added consisting of eligible participants with Parkinson's Disease (Part C).

In Part C (MAD with Parkinson's Disease) eligible PD participants will arrive the evening before initiation of study drug dosing. No Parkinsonism medications will be given after midnight, the following morning potential participants will be clinically assessed in the practically-defined OFF state using MDS-UPDRS Part III. Cohorts will consist of eight (8) subjects, six (6) of whom will receive treatment with IkT-148009 and two (2) with matching placebo daily for up to seven consecutive days. Subjects in each cohort will be observed for 48 hours after their last dose before deciding to initiate the next (higher dose) cohort. Each cohort will be dosed at approximately weekly intervals in order to allow adequate time for collection and review of safety and PK data.

ELIGIBILITY:
Inclusion Criteria Parts A, B:

* 1. Subject must have all questions about the study answered and must have signed the informed consent document before any study-specific procedures are performed.

  2. Men or women aged 55 to 70 years (both inclusive) of any race. 3. Subjects must be otherwise healthy and ambulatory, with no history or evidence of clinically relevant medical disorders as determined by the Investigator in consultation with the Sponsor.

  4. Mini Mental State Examination (MMSE) ≥ 28 at Screening (V1) and Baseline (V2).

  5. Physical examination, clinical laboratory values, vital signs (as defined in the CRU standard operating procedure [SOP]), and the electrocardiogram (ECGs) are clinically acceptable to the Investigator. Body weight ≥ 45 kg at screening and baseline visits. Body Mass Index (BMI) ≥ 18 and ≤30 kg/m2 at screening.

  6. Female subjects must be postmenopausal (12 months without menses and confirmed by follicle stimulating hormone [FSH] > 40 mIU/mL) or surgically sterile (hysterectomy or bilateral oophorectomy) or sterile for other medical reason (i.e., able to document premature low ovarian reserve, birth defect, other). Women who are several years postmenopausal may be considered for enrollment even with [FSH] below this threshold.

  7. Male subjects must agree to practice an acceptable method of highly effective birth control from the Screening visit, while on study and for 7 days after receiving the last dose of study drug. Highly effective methods of birth control include sexual abstinence; vasectomy; or a condom with spermicide (men) in combination with their partner's highly effective method.

  8. Males must be willing to abstain from sperm donation from the screening visit, while on study and through 30 days after receiving the last dose of study drug.

Part C:

Participants must be eligible as in Part A and B, with the following differences/additions:

9. MMSE ≥ 26 at screening (V1) and Baseline (V2) 10. Diagnosis of Parkinson's Disease (consistent with the UK PD Society Brain Bank Criteria for the Diagnosis of PD), with bradykinesia and a clear motor response to levodopa.

11. Hoehn & Yahr staging of 3 or less in the ON state. 12. Good clinical response to levodopa as judged by participant and investigator.

13. Stable doses of all PD medications for at least 4 weeks prior to Screening. 14. Approved by an Enrollment Authorization Committee (EAC).

Exclusion Criteria Parts A and B:

* 1. Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at the screening and admission visits. Abnormalities considered to be non-clinically significant by the Investigator are acceptable.

  2. Clinically significant abnormal findings on physical examination or 12-lead electrocardiogram (ECG) at the screening or admission visits. NOTE: QTcF interval of > 450 msec in males or > 470 msec in females will be the basis for exclusion from the study. Safety ECG may be repeated for confirmatory purposes if initial values obtained exceed the limits specified.

  3. Significant history (within six months prior to receiving the study drug) and/or presence of clinically significant medical, surgical or psychiatric disorder. Subjects with co-morbid conditions that are stable and controlled may remain eligible (stable defined as no change in the dose or frequency of medications over the prior three months).

  4. For optional lumbar puncture: participants with bleeding disorders, relevant lab abnormalities (Screening INR greater than 1.4, platelets less than 50), relevant blood dyscrasias, prior intolerance of LP, anatomical reasons preventing safe or successful collection of fluid (skin infection at site of puncture, relevant spine surgery, spinal deformity, etc), known intracranial space-occupying lesions with mass effect, posterior fossa masses, or relevant brain malformations (Arnold-Chiari malformation, etc), exam findings suggestive of increased intracranial pressure, or known allergy/sensitivity to lidocaine or its derivatives will not be eligible.

  5. eGFR < 60 mL/min 6. Creatinine, Amylase and/or Lipase > ULN 7. Any malignancy in the 5 years prior to screening excluding basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated.

  8. Any subject with a history, presence and/or current evidence of serologic positive result for hepatitis B surface antigen, hepatitis C antibodies, or HIV antibodies 1 or 2. Subjects considered to be cured for hepatitis C will be eligible. 9. Recent history (within previous six months prior to screening) of alcohol or drug abuse (as judged by the investigator) or has consumed > 2 alcohol drinks/day during the last three months prior to screening (one glass is approximately equivalent to: beer [284 mL], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]). Subjects that consume three glasses of alcoholic beverages per day but less than 14 glasses per week may be enrolled at the discretion of the Investigator. Positive screens for alcohol or controlled substances at the screening or admission visits will disqualify a subject from study participation.

  10. Any subject with known hypersensitivity to IkT-148009.

  11. Donation of blood or acute loss of blood within 60 days prior to screening visit.

  12. Any subject who has received treatment with an investigational drug during the 30 days prior to screening.

  13. Investigative site personnel or their immediate families (spouse, parent, child or sibling whether biological or legally adopted).

  14. Any subject unwilling or unable to comply with study procedures.

and in addition for Part C:

15. For optional lumbar puncture: participants with bleeding disorders, relevant lab abnormalities (Screening INR greater than 1.4, platelets less than 50), prior intolerance of LP, anatomical reasons preventing safe or successful collection of fluid (skin infection at site of puncture, relevant spine surgery, spinal deformity, etc), known intracranial space-occupying lesions with mass effect, posterior fossa masses, or relevant brain malformations (Arnold-Chiari malformation, etc), exam findings suggestive of increased intracranial pressure, or known allergy/sensitivity to lidocaine or its derivatives will not be eligible.

16. Diagnosis of secondary or atypical parkinsonism 17. Prior neurosurgery for PD or treatment with DUODOPA or infused apomorphine 18. Concurrent use of neuroleptic medications or other dopamine antagonists. 19. Severe or disabling fluctuations or dyskinesias that would, in the opinion of the investigator, interfere with completion of the study 20. Clinically significant hallucinations or delusions that, in the opinion of the investigator or EAC, may preclude completion of the study 21. Clinically significant orthostatic hypotension that, in the opinion of the investigator, may preclude completion of the study 22. Currently active major depression as determined by BDI-II score of >19 23. Previous surgical procedure for PD.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of abnormal vital sign measurements | Safety assessments performed from Day 1 through Day 14
  body temperature by mouth, blood pressure, pulse rate, pulse oximetry, respiration rate
Safety: incidence of abnormal Clinical Laboratory Data | Safety assessments performed from Day 1 through Day 14
  Clinical chemistry tests will include albumin, alkaline phosphatase, total bilirubin, calcium, cholesterol, creatinine, creatinine clearance, creatinine kinase (CK), gamma-glutamyltransferase (γ-GT), glucose, lactate dehydrogenase (LDH), inorganic phosphorus, lipase, amylase, potassium, magnesium, total protein, aspartate transaminase (AST), alanine transaminase (ALT), sodium, triglycerides, urea and uric acid, bicarbonate and chloride. TSH levels will also be monitored. CBC assessments will include hemoglobin, hematocrit, red blood cell (RBC) count, reticulocyte count, white blood cells (WBC) count with differential, platelet count and PT-INR. PT-INR should be reported in both prothrombin time and international normalized ratio. Men and women will undergo additional laboratory tests for reproductive organ function to include leutenizing hormone (LH), follicle stimulating hormone (FSH), testosterone and inhibin B.
Safety: incidence of abnormal electrocardiogram [ECG] | Safety assessments performed from Day 1 through Day 14
  An ECG traces the electrical activity of the heart.
Safety: C-SSRS | Safety assessments performed from Day 1 through Day 14
  Columbia Suicide Severity Rating Scale questionaire
Tolerability (adverse event reporting) | Day 1 through 14 days post last dose
  Adverse events reported
Pharmacokinetic AUC of IkT-148009 | Part A: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post dose. Part B: As in Part A plus 120, 144, 168, 192 hours post-dose.
  Area under the concentration-time curve (AUC0-∞)
Pharmacokinetic Cmax of IkT-148009 | Part A: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post dose. Part B: As in Part A plus 120, 144, 168, 192 hours post-dose.
  Maximum plasma concentration (Cmax)
Pharmacokinetic AUC to last time point of IkT-148009 | Part A: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post dose. Part B: As in Part A plus 120, 144, 168, 192 hours post-dose.
  Area under the concentration-time curve from time zero to last time point (AUC0-last)
Pharmacokinetic Tmax of IkT-148009 | Part A: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post dose. Part B: As in Part A plus 120, 144, 168, 192 hours post-dose.
  Time to reach maximum concentration (Tmax)
Pharmacokinetic distribution half-life of IkT-148009 | Part A: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post dose. Part B: As in Part A plus 120, 144, 168, 192 hours post-dose.
  The distributional half-life and terminal half-life (t1/2)
Pharmacokinetic trough concentration of IkT-148009 | Part A: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours post dose. Part B: As in Part A plus 120, 144, 168, 192 hours post-dose.
  Exposure (Ctrough)
Pharmacokinetic concentration of IkT-148009 steady-state at maximum concentration | Part B, C: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192 hours post-dose.
  Exposure (Cmax SS)
Pharmacokinetic exposure of IkT-148009 steady-state | Part B, C: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192 hours post-dose.
  Exposure (AUC SS)

OTHER OUTCOMES:
Exploratory Biomarker Screen of protein factors | Part B and C only, up to 1 year
  Biomarker screen in CNS-derived exosomes
Exploratory Biomarker Screen of drug concentration | Part B and C only, up to 1 year
  IkT-148009 drug concentrations in the CSF in Parts B, C portion of this study only.
Change from Baseline to Final visit in the MDS-UPDRS Motor Subscale (Part III) Score | Part C only, up to 1 year
  MDS-UPDRS motor subscale
Change from Baseline to Final Visit in the MDS-UPDRS Non-motor aspects of experiences of daily living (Part I) Score and in the MDS- UPDRS Motor aspects of experiences of daily living (Part II) Score. | Part C only, up to 1 year
  MDS-UPDRS Parts I + II subscale
Clinical Global Impression of Improvement (CGI-I) Score and the Patient Global Impression of Change (PGI-C) Score between Baseline and Final visit | Part C only, up to 1 year
  CGI-I score
Change in Non-Motor Symptom Score (NMSS) | Part C only, up to 1 year
  NMSS score
Change from Baseline to Final Visit in Parkinson's Disease Questionnaire 39 (PDQ-39). | Part C only, up to 1 year
  PDQ-39 score
Change from Baseline to Final Visit in the Patient Global Impression of Severity Score (PGI-S) | Part C only, up to 1 year
  PGI-S score
Change from Baseline to Final Visit in Complete Bowel Movement Score (CSBM). | Part C only, up to 1 year
  CSBM score
Change in Patient Assessment of Upper GI Disorders Severity Index (PAGI-SYM) | Part C only, up to 1 year
  PAGI-SYM score

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hassman, MD, Principal Investigator — Hassman Research Institute; Larry Blob, MD, Study Chair — Cognitive Research Corporation
Locations (4):
- United States (4):
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Velocity Clinical Research, Hallandale, Florida
  - Quest Research Institute LLC, Farmington Hills, Michigan
  - Hassman Research Institute, Marlton, New Jersey